CLINICAL TRIAL: NCT03236363
Title: Effectiveness of MOVI Interventions on Improving Adiposity, Cognition and Motor Competence by Increasing Aerobic Cardiorespiratory Fitness: MOVI-da10!
Brief Title: Effectiveness of MOVI Interventions on Adiposity, Cognition and Motor Competence: MOVI-da10!
Acronym: MOVI-da10!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI16b/01919
Record Dates: First submitted 2017-07-21; First posted 2017-08-01 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity; Children; Obesity; Cardiovascular; Cardiorespiratory Fitness
Keywords: Physical activity; Obesity; Children; Cognitive function; Academic achievement; Cardiorespiratory fitness; Adiposity; Cardiovascular fitness; Aerobic capacity
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MOVI-da 10! active breaks (Experimental): It is a physical activity intervention that consists on two daily physical activity active breaks of 10 minutes of duration (intensity: 4-6 METs, Heart rate ≥150 bpm). It is aimed to enhance physical activity, motor skills and cognition among 5 years old children
  Interventions: Behavioral: MOVI-da10! active breaks
- Control (No Intervention): No intervention
- MOVI-da10! integrated physical activity (Experimental): It is an integrated physical activity intervention that consists on two daily cognitive demanding physical activity breaks of 10 minutes of duration (intensity: 2-3 METs, Heart rate <150 bpm). It is aimed to enhance physical activity, motor skills and cognition among 5 years old children
  Interventions: Behavioral: MOVI-da10! integrated physical activity

INTERVENTIONS:
Behavioral: MOVI-da10! active breaks — MOVI-da10! active breaks, is a physical activity intervention that consists on two daily physical activity breaks of 10 minutes of duration (intensity: 4-6 METs, Heart rate ≥150 bpm). It is aimed to enhance physical activity, motor skills and cognition among 5 years old children
  Arms: MOVI-da 10! active breaks
Behavioral: MOVI-da10! integrated physical activity — MOVI-da10! integrated lessons, is a physical activity intervention that consists on two daily cognitive demanding physical activity breaks of 10 minutes of duration (intensity: 2-3 METs, Heart rate <150 bpm). It is aimed to enhance physical activity, motor skills and cognition among 5 years old children
  Arms: MOVI-da10! integrated physical activity

SUMMARY:
Project which objective is to test the effectiveness of a classroom-based physical activity intervention (MOVI-da10!) on improving, body composition, cardio-respiratory fitness and executive function.

DETAILED DESCRIPTION:
In the last decade, this research group has tested the effectiveness of three interventions following after-school intervention model. The first one (MOVI) was carried out in peripuberal age children (4th and 5th year of primary education, 8-11 years) and showed a moderate effect in reducing the adiposity of schoolchildren with higher BMI, an improvement of the lipid profile, without significantly improving the global cardiometabolic risk because it did not produce a reduction in insulinemia.

The second edition (MOVI-2), carried out at schoolchildren of the same age range, increased the duration and intensity of the sessions, and was focused on the development of muscular strength in order to improve insulinemia levels. The intervention showed proved effectiveness; in addition, the data from this intervention showed a modest improvement in girls' aerobic capacity, but not in boys.

The last edition (MOVI-KIDS) was aimed at children aged 4 to 7 years to test the hypotheses that vigorous physical activity at early ages could produce lifelong cardio-metabolic benefits. Data submitted for publication in this study show that, as in the case of the IDEFICS study in children of similar age, the intervention was not effective in improving fitness.

This new edition (MOVI-da10!) has been designed following integrated physical activity intervention and active breaks designs, and as a controlled cluster-randomized trial including 9 schools from Cuenca province, Spain. Six schools will be randomized to the two intervention groups (IG), where the intervention of MOVI-da10! will be conducted for third grade preschool children (about 5 years old), using two different design. Three of them will receive an active breaks intervention, in which twice a day a 10 minutes breaks standard physical activity will be developed, and the other three will receive twice a day a 10 minutes of enriched physical activity integrated in the curriculum. The other three schools will be allocated to the control group (CG).

During an academic year the MOVIda10! interventions will consist of: i) an integrated across the curriculum cognitive demanding physical activity program including two active breaks lasting 10 min, five days/week; and ii) an active breaks physical activity program including two active breaks lasting 10 min, five days/week. In the CG regular physical activity will continue.

At the end of the school year the researchers will determine main outcome variables: changes in VO2max, body fat by bioimpedance and executive function.

The hypotheses of this new edition will be that: the MOVI-da10 intervention! based on physical activity integrated in the curriculum for third grade preschool children, will be:

1. Moderately increase the executive function and academic performance in the IGs versus the CG (effect size 0.5).
2. Increase aerobic capacity (VO2max) in IGs versus CG by 3%.
3. Reduced body fat in IGs versus CG by 3%

ELIGIBILITY:
Inclusion Criteria:

* Schools must have at least one full classrooms for the 3rd year of preschool.
* The approval of boards of governors will be necessary to participate in the intervention and in the measurements at the beginning and end of academic year.
* Children's parents or legal representatives will sign an informed consent to participate.
* Children's parents will be invited to collaborate by filling in questionnaires with regard to family leisure habits, sleeping, eating and getting around town.

Exclusion Criteria:

* Children with severe Spanish language learning difficulties.
* Children with serious physical or mental disorders identified by parents or teachers that would impede participation in the programme's activities
* Children diagnoses of chronic disorders, such as heart disease, diabetes or asthma, which in the opinion of their paediatricians would prevent their participation in the programme's activities (MOVI-da10!).

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Executive function | One year
  Executive function will be measured by standardized test using the NIH toolbox

SECONDARY OUTCOMES:
VO2 max | One year
  It will be assessed by using 20-m shuttle run test, which is validated to measure maximal aerobic capacity in children.
Motor skills | One year
  By using the Movement Assessment Battery for Children 2 (M-ABC 2)
Body fat% | One year
  Body fat percentage measured by Bioimpedance analysis
Health-related quality of life | One year
  By using the validated version in Spanish of KIDL for children of 4-7 years and their parents.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Martinez-Vizcaino, PhD, MD, Principal Investigator — Social and Health Care Research Center, University of Castilla-La Mancha
Locations (1):
- Social and Health Research Center. Universidad de Castilla-La Mancha, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Lopez M, Ruiz-Hermosa A, Redondo-Tebar A, Visier-Alfonso ME, Jimenez-Lopez E, Martinez-Andres M, Solera-Martinez M, Soriano-Cano A, Martinez-Vizcaino V; MOVI group. Rationale and methods of the MOVI-da10! Study -a cluster-randomized controlled trial of the impact of classroom-based physical activity programs on children's adiposity, cognition and motor competence. BMC Public Health. 2019 Apr 18;19(1):417. doi: 10.1186/s12889-019-6742-0. PMID 30999870